CLINICAL TRIAL: NCT04444323
Title: 3D Telemedicine During COVID-19: Cohort Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: Jean Brown Bequest Fund, Glasgow (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GN20HS300
Record Dates: First submitted 2020-06-20; First posted 2020-06-23 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Telemedicine; Surgery, Plastic
Keywords: 3-D

STUDY DESIGN:
Intervention Model Description: Single cohort patients seen face-to-face and then by 3D telemedicine
Masking Description: Data analysis will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D Telemedicine (Experimental): Single arm. All patient seen face-to-face and then with 3D telemedicine.
  Interventions: Other: 3D Telemedicine

INTERVENTIONS:
Other: 3D Telemedicine — The intervention is a consultation conducted using a 3D form of telemedicine

SUMMARY:
It is critical to establish an effective form of telemedicine during the Covid 19 pandemic, that will allow safe social distancing of clinicians and patients. Canniesburn Regional Plastic Surgery and Burns Unit serves as the regional plastic, burns and reconstructive centre for West of Scotland, population 3 million. All face to face clinics have been cancelled and converted to telephone/telemedicine only consultations. The research will establish both 2D and 3D telemedicine as normal patient follow up practice during this period.The project therefore aims to implement a 3D telemedicine system to facilitate patient follow up and remote physiotherapy, that will act as if the patient is physically 'present' in the room. Physiotherapy is crucial to patient outcomes after burns contractures, hand trauma and cancer reconstruction. The 3D telemedicine system will be built by an industrial partner, with CE marked equipment, specifically to help during the Covid-19 Pandemic.

DETAILED DESCRIPTION:
1. Background:

   Telemedicine is critical during Covid pandemic. A seismic shift in clinical practice has occurred in the UK, with nearly all medical clinics cancelled or converted to telephone or telemedicine clinics (Attend Anywhere or Zoom). These fail to adequately substitute for a face-to-face consultation, with the National Health Service (NHS) needing higher quality, more clinically effective methods of remote patient interaction. This project will be the world's first evaluation of a novel, potentially transformative form of 3D telemedicine, facilitating telepresence as if the patient were in the room. This state-of-the-art system has been developed by an industrial partner, specifically to help with remote patient communication during Covid pandemic. This uses an array of 3D cameras connected to fusion and render servers, allowing reconstruction of a 3D image in real time. This may give more information about a patient's condition, particularly in more visual specialties such as Plastic Surgery

   The research will fulfil criteria for the European Commission's Model for Assessment of Telemedicine applications (MAST, Kidholm 2012). This will include participatory design, and evaluation with a preliminary cohort study, to shape the follow on research. This will assess clinicians' and patients' perception of system usability, delivery of therapies, clinical accuracy and interaction. On project completion, fulfilment of MAST criteria will enable upscaling and lead onto a randomized trial. The study design will be informed by participatory design prior to the start of the clinical study. This will include clinical stakeholders (specialist nurses, doctors and physiotherapists), the digital research team, and patient groups. The focus groups will collate user groups opinions about the 3D system, functionality, risks, and applicability.

   The clinical study will be a feasibility study involving clinician and patient feedback on 3D telemedicine, and will additionally collect safety, reliability and fidelity data. The study will be a mixed methods analysis assessing measures of usability, satisfaction, presence, task load index, and accuracy. Clinicians and patients will complete questionnaires and undergo a short interview on the use of both forms of telemedicine. There are no data regarding the use of 3D telemedicine, but this will leverage study design and validated questionnaires from other similar studies (Buvik 2016). The study will continue as post covid services are being established.
2. Aims

   This study will refine and pilot the feasibility of introducing 3D telemedicine into plastic surgery clinics and gain pilot data on the comparative efficacy and acceptability compared to face-to-face clinics, from both a patient and clinician perspective. The feasibility study will then inform the design and size of larger randomised study to compare 2D and 3D telemedicine.
3. Research Questions Primary

   • Understand the feasibility and acceptability of introducing 3D telemedicine into plastic surgery clinics, in particular assessing safety, reliability and feedback data.

   Secondary
   * Provide preliminary evidence regarding how 3D telemedicine compares to face-to-face consultations using clinician and patient assessments
   * Assess the appropriate rating scales/instruments to take forward to a RCT
   * Provide preliminary objective data to assess the accuracy of 3D telemedicine to determine clinical measurements (where applicable e.g. angles of contracture in hand) and outcome scoring scales (where applicable e.g. validated Unilateral Cleft Score Surgical Outcomes Evaluation Scale - UCLSOE)
   * Provide preliminary data for machine learning training to Strathclyde University
   * Safety and reliability measures of the system (number of failed and interrupted 3D telemedicine consultations).
   * To assess if clinical outcomes determined by 3D Telemedicine are similar to face-to-face
4. Study Design

Pre-study protocol optimisation will include data from a patient feedback study and a clinician feedback study. This will provide feedback for incremental system improvement and baseline outcome data. This will be followed by a Clinician Cohort Trial.

4A. Patient Feedback Study

Focus groups will co-design the features and functionality of the 3D Telemedicine, and inform clinical/patient feedback questionnaires. Clinical stakeholders (specialist nurses, doctors and physiotherapists), the digital research team and patient groups (existing user groups in breast cancer, sarcoma, cleft, hand surgery and physiotherapy) will be invited to participate in focus groups. The discussion will explore user groups opinions and ideas about the 3D system, functions that they would like to see implemented, and scenarios where this may be advantageous over a standard 2D system, and potential risks, using open ended questions. The patient group will consist of 40 patients sampled from existing user groups and will include patients already known to the research team. These patients will be invited to participate in a feedback study and will be examined by both 3D and 2D Telemedicine by their usual care clinician, and without any randomisation. They will be then asked to complete a feedback questionnaire and interview. Patient outcomes assessed will include:

Satisfaction: Visual Analogue Scale 0-100 Mental Effort Rating Scale - single instrument Likert scale (Paas 1996) System Usability Scale - 10 item industry standard technology scale Single Item Presence Questionnaire - This will ask patients the question "To which extent did you feel present in the virtual clinic, as if you were really there?". This is a single item evaluation of presence validated by Bouchard et al 2004.

Telehealth Usability Questionnaire - 21 item scale - assessment of telemedicine (TUQ, Parmanto 2016) Semi Structured exit interview - will discuss with participant their views on the telemedicine system, using "Keep, Lose and Change" feedback prompts to help in incremental system improvements.

4B. Clinician Feedback Study

A group of 25 clinicians including nurses, doctors and physiotherapists, will be invited to assess both 3D and 2D Telemedicine systems without randomisation, with a member of the research team acting as a "patient". They will be then asked to complete a feedback questionnaire and interview. Clinician outcomes assessed will include:

Satisfaction: Visual Analogue Scale 0-100 Mental Effort Rating Scale - single instrument Likert scale (Paas 1996) System Usability Scale - 10 item industry standard technology scale Presence Questionnaire - 29 item scale - assessment of presence in the system/virtual environment (PQ, Witmer 2005).

Telehealth Usability Questionnaire - 21 item scale - assessment of telemedicine (TUQ, Parmanto 2016) Semi Structured exit interview - will discuss with participant their views on the telemedicine system, using "Keep, Lose and Change" feedback prompts to help in incremental system improvements.

4C. Cohort Study

Patient Identification Patients will be recruited for this study from plastic surgery clinics, including breast cancer, sarcoma, head & neck reconstruction, flap reconstruction, limb reconstruction, hand trauma, burns and cleft lip. Clinicians recruited to the study be from Canniesburn Regional Plastic Surgery and Burns Unit. The wide spectrum of clinical cases including in this cohort trial will allow increased generalizability of the results.

Inclusion criteria

* Patients 1-95 years old (children will include post-cleft lip repair)
* Patients able to read and understand English
* Patients able to give informed consent

Exclusion criteria

* Patients not meeting the inclusion criteria
* Patients who do not have capacity to consent
* Patients who are registered blind or deaf

Consent The patient information sheets (PIS) will be sent to the patients for their consideration prior to them attending their clinic appointment. The nurse will then take the patient into a private telemedicine clinic room to go through the PIS with them and answer any questions. If the patient wishes to participate, the nurse will provide a consent form which has some statements to agree to and sign. The patient can keep a copy of the signed consent form as well as the PIS.

Additional consent will be taken for opting into photo or video recordings. Telemedicine data may be used in further research, including machine learning. The PIS will make it clear to the patient that a copy of their identifiable images will be held for research purposes.

The PIS and consent will also explain that the our industrial partner will have access to the data, system and images (covered by a data processing agreement and 3rd Party Access agreement) to resolve any image quality, render, fusion, or transmission problems.

Study procedures

All patients will be assessed first face-to-face, and subsequently with 3D telemedicine by a separate clinician. In addition to the standard consultation, all patients will have the range of motion of the right and left elbows measured face-to-face with blinded (scales hidden) goniometers, and on the 3D system with a blinded on-screen goniometer. Patients will fill in a questionnaire and undertake a short exit interview after completion of consultations. Clinicians involved in this study will be asked to fill in a clinician consent form, and will be provided with a clinician information sheet prior to the study. The clinician fills in a questionnaire on the use of telemedicine for each patient, and undergoes an exit interview just once at the end of the study. The data for the elbow range of motion will be stored on computer and the clinician will re-measure at 1 week (patient does not need to return).

The Clinician telemedicine questionnaire will be filled in once per patient and comprises 71 items from the following rating scales.

Mental Effort Rating Scale - single instrument Likert scale (Paas 1996) University of North Northway - 5 item - telemedicine questionnaire (UNN, Buvik 2016) System Usability Scale - 10 item industry standard technology scale Presence Questionnaire - 29 item scale - assessment of presence in the system/virtual environment (PQ, Witmer 2005).

Telehealth Usability Questionnaire - 21 item scale - assessment of telemedicine (TUQ, Parmanto 2016) NASA task load index (NASA TLX) - 5 item modified scale - an indication of the ease of performing a task and frustration levels.

Semi Structured exit interview - will discuss with participant their views on the telemedicine system, what went well, and what can be improved.

The clinician conducting the face-to-face will complete a shortened questionnaire with the UNN scale only. The patient will fill also fill in a shortened questionnaire with a maximum of 37 items, including the Mental Effort Rating Scale, Telehealth Usability Questionnaire, NASA TLX and System Usability Scale.

The telemedicine consultation will include clinical outcome scales (where applicable e.g. unilateral cleft outcome scoring) recorded as part of normal practice. This will be compared to actual clinical outcomes taken in clinic on the same day (to provide "ground truth" for comparison with telemedicine measurements).

Safety and reliability data will be collected throughout the study, incuding:

1. Failed 3D telemedicine visits - failure and interruption, including reasons e.g. network/ software/ hardware. In event of failure a face to face consultation will still take place.
2. Image aberration - record of subjective distortion/ noise.
3. Correlation of face-to-face and telemedicine patient outcomes and findings

The 3D system will be permanently set up in a locked clinic room in a non-covid hospital. The system can be switched to 2D if required.

The 3D telemedicine system will comprise:

* 80/20 aluminium frame support for cameras
* 8 3D cameras
* 2 Patient LED screens
* Fusion and render computers
* At 'receiving' end - standard computer and LED screen

The system will be simple to use - 3D images will be viewed on a screen and can be manipulated in space, enlarged, and frozen using mouse controls. The research team's industrial partner will have provided training of clinic staff on how to operate the equipment and support of the equipment during the data collection activity. Training of the participating clinicians will take the form of a short introductory session by the research team at the start of each research clinic. The patient will likewise be shown how to use the system, but there will be no need for the patient to use any controls or interface.

Follow Up

There is no follow up required - patients are only required to attend an extended clinic visit and complete the study questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast cancer reconstruction
* Patients with sarcoma
* Patients with head & neck reconstruction
* Patients with flap reconstruction
* Patients with limb reconstruction
* Patients with hand trauma
* Patients with burns
* Patients with cleft lip
* Patients able to read and understand English
* Patients able to give informed consent

Exclusion Criteria:

* Patients not meeting the inclusion criteria
* Patients who do not have capacity to consent
* Patients who are registered blind or deaf

Ages: 1 Year to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-07-10 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Presence Questionnaire | Single time point at day 1 (Clinician assesses telemedicine system once after seeing patient) ]
  Version 3 of PQ, 29 item rating scale of "presence". Witmer 2005

SECONDARY OUTCOMES:
University Hospital of North Northway Questionnaire | Single time point at day 1 (Clinician assesses telemedicine system once after seeing patient) ]
  5 item questionnaire on telemedicine quality. UNN Buvik 2016.
Telehealth Usability Questionnaire | Single time point at day 1 (Clinician assesses telemedicine system once after seeing patient) ]
  21 item scale - assessment of telemedicine (TUQ, Parmanto 2016)
System Usability Scale | Single time point at day 1 (Clinician assesses telemedicine system once after seeing patient) ]
  10 item industry standard technology scale
Mental Effort Rating Scale | Single time point at day 1 (Clinician assesses telemedicine system once after seeing patient) ]
  Single instrument Likert scale (Paas 1996)
NASA TLX | Single time point at day 1 (Clinician assesses telemedicine system once after seeing patient) ]
  Measure of task load index - 5 item modified scale - an indication of the ease of performing a task and frustration levels.
Range of Motion measurements for elbow joint | Single time point at day 1 (Clinician assesses telemedicine system once after seeing patient) ]
  Range of Motion measurements for elbow joint measured with face-to-face goniometer or on computer (telemedicine)

OTHER OUTCOMES:
Reliability | Single time point at day 1 (whether telemedicine is successful)
  Proportion of completed, successful telemedicine consultations
Image distortion | Single time point at day 1 (whether telemedicine has distortion)
  Proportion of telemedicine consultations suffering image quality distortion

CONTACTS AND LOCATIONS:
Locations (1):
- Canniesburn Regional Plastic Surgery and Burns Unit, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share data

REFERENCES:
- [Derived] Lo S, Fowers S, Darko K, Spina T, Graham C, Britto A, Rose A, Tittsworth D, McIntyre A, O'Dowd C, Maguire R, Chang W, Young D, Hoak A, Young R, Dunlop M, Ankrah L, Messow M, Ampomah O, Cutler B; 3DTM (3D Telemedicine) Collaborative research group; Armstrong R, Lalwani R, Davison R, Bagnall S, Hudson W, Shepperd M, Johnson J. Participatory development of a 3D telemedicine system during COVID: The future of remote consultations. J Plast Reconstr Aesthet Surg. 2023 Dec;87:479-490. doi: 10.1016/j.bjps.2022.10.012. Epub 2022 Oct 13. PMID 36890078